CLINICAL TRIAL: NCT01169038
Title: Investigation of the Efficacy of Antibiotics on Pulmonary Sarcoidosis
Acronym: CLEAR Lung
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Wonder Drake, Associate Professor of Medicine, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 100552
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Pulmonary Sarcoidosis; Lung Function
Keywords: sarcoidosis; mycobacteria; lung; pulmonary; radiographic improvement
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis; Mycobacterium Infections | interventions — Levofloxacin; Ethambutol; Rifampin; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Antibiotics (Active Comparator): Levaquin 750 mg loading on day 1, then 500 mg po QD Ethambutol 15-25 mg/kg for a maximum of 1200mg po QD Azithromycin 500mg on day 1, then 250 mg po QD
  **Rifampin 10 mg/kg for a maximum of 600mg po QD or Rifabutin 10 mg/kg for a maximum of 300 mg po QD. **We will not use both, but either one or the other based upon if the patient is on other medications that are metabolized by the cytochrome P450 pathway.
  Interventions: Drug: levaquin; ethambutol; rifampin and azithromycin.

INTERVENTIONS:
Drug: levaquin; ethambutol; rifampin and azithromycin. — Levaquin 750 mg loading on day 1, then 500 mg po QD Ethambutol 15-25 mg/kg for a maximum of 1200mg po QD Azithromycin 500mg on day 1, then 250 mg po QD
  **Rifampin 10 mg/kg for a maximum of 600mg po QD or Rifabutin 10 mg/kg for a maximum of 300 mg po QD. **We will not use both, but either one or the other based upon if the patient is on other medications that are metabolized by the cytochrome P450 pathway.

SUMMARY:
Sarcoidosis is a granulomatous disease for which the molecular and immunologic association with mycobacteria continues to strengthen. The investigators are interested in conducting a proof-of-concept investigation of the effects of antibiotics on sarcoidosis resolution. The investigators hypothesize that pulmonary sarcoidosis will improve faster if patients are given antimycobacterial therapy, in addition to their standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with sarcoidosis will be enrolled as defined below.

  1. Patients with sarcoidosis as defined by the ATS/ERS/WASOG statement on sarcoidosis as defined by the clinical presentation consistent with sarcoidosis, as well as biopsy finding granulomas, and no alternative for the cause of the granulomas, such as tuberculosis.
  2. Evidence of parenchymal disease on chest radiograph (Stage II, III or IV) or Stage I disease by chest radiographs and evidence of abnormal spirometry. . Subjects with concurrent extrapulmonary sarcoidosis, particularly skin and eye involvement, can be enrolled.
  3. FVC of >=45% and <=80% of predicted normal value at screening.
  4. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy), or is using one of the following methods of birth control for the duration of the study and 90 days after study completion:

     1. condoms, sponge, foams, jellies, diaphragm, or intrauterine device
     2. contraceptives (oral or parenteral) for three months prior to study drug administration
     3. a vasectomized sole partner
     4. Females of childbearing potential must have a negative urine pregnancy test at screening visit.

Exclusion Criteria:

* 1. No consent/inability to obtain consent. 2. Age less than 18 years of age. 3. Inability to draw blood. 4. ALT or AST >5 times upper limit of normal (ULN) 5. Pregnancy or breast feeding. 6. Allergy to macrolides, quinolones or rifamycins. 7. Visual Impairment as defined by differentiating colors per personal history. 8. Family or personal history of long QT syndromes. 9. Patients receiving another interventional investigational drug for sarcoidosis within the 30 days prior to dosing 10. Use of any investigational medication within the past 28 days prior to study enrollment.

  11. Subject has been hospitalized for infection or received IV antibiotics within the previous 2 months prior to baseline.

  12. Subject has a history of tuberculosis at anytime or close contact with a person with active tuberculosis within the previous 6 months, or persistent or active infections requiring hospitalization or treatment with IV antibiotics, IV antiretrovirals, or IV antifungals within 30 days of baseline, OR oral antibiotics, antivirals, or antifungals for purpose of treating infection, within 14 days of baseline.

  13. Subject has an active infection requiring systemic antibiotics at time of screening 14. Subject has a history of listeriosis, treated or untreated tuberculosis, exposure to individuals with tuberculosis.

  15. Have a diagnosis of other significant respiratory disorder other than sarcoidosis that would complicate the evaluation of response to treatment 16. Patients otherwise unsuitable for participation in the opinion of the investigator.

  17. No smoking for past one year.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wonder P Drake, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University School of Medicine, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Drake WP, Richmond BW, Oswald-Richter K, Yu C, Isom JM, Worrell JA, Shipley GR. Effects of broad-spectrum antimycobacterial therapy on chronic pulmonary sarcoidosis. Sarcoidosis Vasc Diffuse Lung Dis. 2013 Nov 25;30(3):201-11. PMID 24284293

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from outpatient pulmonary clinics at Vanderbilt University Medical Center and the surrounding community between July 14 and August 24, 2010. All patients met American Thoracic Society/European Respiratory Society/World Association of Sarcoidosis and Other Granulomatous Diseases (ATS/ERS/WASOG) criteria.
Period: Overall Study
Arm/Group | Antibiotics
Started | 15
Completed | 8
Not Completed | 7
Not completed — Death | 1
Not completed — Adverse Event | 5
Not completed — Required antibiotic administration | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antibiotics
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 54 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Absolute FVC From Baseline to Post Completion of 8 Weeks of Antibiotic Therapy.
Description: The primary endpoint was improvement in absolute FVC from baseline to completion of therapy. Spirometry testing was performed using a standardized calibrated laptop spirometer, Flowscreen II USA Spirometer (VIASYS Healthcare Inc., Yorba Linda, CA). The volume accuracy of the spirometer was checked daily using a three liter calibration syringe. Each subject was given at least three attempts and the greatest measurement for absolute FVC and Forced Expiratory Volume (FEV1) at baseline, four week, and eight week assessments was recorded.
Time Frame: 8 weeks
Population: In the ITT analysis, we included the values from the last measured value for those who did not complete the trial. We analyzed the measured value at 8 weeks among those subjects who completed 8 weeks of therapy in the per protocol analysis.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Antibiotics
Number analyzed (Participants) | 15
liters | 2.61 (1.01)

ADVERSE EVENTS:
Time Frame: The AE were collected over six months.
Arm/Group | Antibiotics
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 8/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antibiotics (N=15)
Arthalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Insomnia (General disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
leucopenia (Blood and lymphatic system disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No